CLINICAL TRIAL: NCT06461975
Title: Effect of Benoxinate Hydrochloride Eye Drops on The Premature Infant Pain Profile Score During Retinopathy of Prematurity Screening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Islam Shereen Hamdy, Associate Professor, Alexandria University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Benoxinate drops for ROP exam
Record Dates: First submitted 2024-06-06; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Retinopathy of Prematurity
Keywords: Infant stress; Retinopathy of prematurity; Benoxinate hydrochloride; PIPP score
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — benoxinate; Lubricant Eye Drops; Hyaluronic Acid; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Prospective, observational, double-blinded, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A dedicated clinical pharmacist placed the topical benoxinate HCL (Benox ®, Removed for facilitating the blinded review). and the artificial tear (Sodium Hyaluronate 2 mg/ml) eye drops (Polyfresh ®, Removed for facilitating the blinded review) in identical bottles, each of them had a code that was changed every clinic and was not known to the examining ophthalmologist, the nurse in charge of swaddling the baby and putting the drops or the attending neonatologist monitoring the infant and recording the PIPP score. The clinical pharmacist would ensure that crossover was performed in the second examination of every study child.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tear substitute in first exam (Experimental): Te first examination was done using the tear substitute eye drops and the second using the Benoxinate HCL drops given just before the ROP screening.
  Interventions: Drug: artificial tear (Sodium Hyaluronate 2 mg/ml) eye drops.
- Benoxinate HCL in first exam (Experimental): infants in Group B had the reversed order of the drops in the two examinations. the first examination done using the Benoxinate HCL drops and the second using the tear substitute eye drops
  Interventions: Drug: Benoxinate Hydrochloride

INTERVENTIONS:
Drug: Benoxinate Hydrochloride — The first group had the first examination done using the tear substitute "Polyfresh ®" eye drops and the second using the Benoxinate HCL drops "Benox ®" given just before the ROP screening.
  Other Names: "Benox ®"
  Arms: Benoxinate HCL in first exam
Drug: artificial tear (Sodium Hyaluronate 2 mg/ml) eye drops. — The second group had the first examination done using the Benoxinate HCL drops "Benox ®" eye drops and the second using the tear substitute "Polyfresh ®"given just before the ROP screening.
  Other Names: "Polyfresh ®"
  Arms: Tear substitute in first exam

SUMMARY:
Aims: To evaluate the effects of topical Benoxinate HCL eye drops on the Premature Infant Pain Profile (PIPP) scores in infants undergoing Retinopathy of Prematurity (ROP) screening.

Methods: A randomized prospective double-masked cross-over trial was conducted on preterm infants screened for ROP at least twice. Dilated fundus examination was done in Group A infants using the tear substitute eye drops and the second using the Benoxinate HCL drops and the reversed order of drops for Group B. Video recording of the pulse oximeter monitor, the face and the body of the infant were analyzed by a single neonatology consultant for Premature Infant Pain Profile (PIPP) scoring 1 minute before, during the examination of the first eye, 1 minute and 5 minutes after the conclusion of the examination of the second eye. The sound of the ophthalmologist on the video recordings indicating the time of the lid speculum insertion, the shining of the indirect ophthalmoscope light without indentation and the scleral indentation would aid in assessing the differences of the PIPP indicators during each step of the examination.

DETAILED DESCRIPTION:
Aims: To evaluate the effects of topical Benoxinate HCL eye drops on Premature Infant Pain Profile (PIPP) scores in infants undergoing Retinopathy of Prematurity (ROP) screening.

Methods: A randomized prospective double-masked cross-over trial was conducted on preterm infants screened for ROP at least twice. Dilated fundus examination was done in Group A infants using the tear substitute eye drops and the second using the Benoxinate HCL drops and the reversed order of drops for Group B. Video recording of the pulse oximeter monitor, the face and the body of the infant were analyzed by a single neonatology consultant for Premature Infant Pain Profile (PIPP) scoring 1 minute before, during the examination of the first eye, 1 minute and 5 minutes after the conclusion of the examination of the second eye. The sound of the ophthalmologist on the video recordings indicating the time of the lid speculum insertion, the shining of the indirect ophthalmoscope light without indentation and the scleral indentation would aid in assessing the differences of the PIPP indicators during each step of the examination.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with GA ≤34 weeks and/or with birth weight ≤2000 g
* Preterm infants with larger GA or birth weight who were at increased risk of ROP according to the attending neonatologist
* Infants were believed to require at least 2 ROP screenings

Exclusion Criteria:

* Infants on muscle relaxants, analgesics, sedatives, or exogenous steroids
* Infants who required mechanical ventilation or continuous positive airway pressure at the first examination

Ages: 28 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
PIPP score | 1-3 month after birth
  The PIPP is a composite measure that includes seven indicators, each of which is rated on a four-point scale (0-3). The indicators include heart rate, oxygen saturation, GA, brow bulge, nasolabial furrow, behavioural state, and eye squeeze. Larger number indicates more stress (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Islam Ahmed, M.D., Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Data are available and owned by the authors and can be shared upon request